CLINICAL TRIAL: NCT01620060
Title: A Phase 1 Open-Label, Multicenter, Single and Multiple Ascending Dose Study to Evaluate Pharmacokinetics, Safety, and Tolerability of Lurasidone in Subjects 6 to 17 Years Old With Schizophrenia Spectrum, Bipolar Spectrum, Autistic Spectrum Disorder, or Other Psychiatric Disorders
Brief Title: Lurasidone Pediatric Pharmacokinetics Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D1050300
Record Dates: First submitted 2012-05-23; First posted 2012-06-15 (Estimated); Results first posted 2014-07-31 (Estimated); Last update posted 2016-04-08 (Estimated); Status verified 2016-03

CONDITIONS: Schizophrenia; Autism
Keywords: Schizophrenia; autism; bipolar; Lurasidone; Latuda
MeSH Terms: conditions — Schizophrenia; Autistic Disorder | interventions — Lurasidone Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lurasidone oral tablets (Experimental): Lurasidone 20, 40, 80, 120 or 160 mg/day
  Interventions: Drug: Lurasidone

INTERVENTIONS:
Drug: Lurasidone — Lurasidone 20, 40,80, 120 or 160 mg/day oral single and multiple does of lurasidone for 12 days

SUMMARY:
This is a Phase 1, open-label, multicenter, single and multiple ascending lurasidone dose study in subjects from 6 to 17 years old with schizophrenia spectrum, bipolar spectrum, autistic spectrum disorder, or other psychiatric disorders.

DETAILED DESCRIPTION:
To characterize lurasidone PK profile following single and multiple oral doses of 20, 40,80, 120 or 160 mg/day lurasidone in the targeted pediatric/adolescent population (6-17 years old)with schizophrenia spectrum, bipolar spectrum, autistic spectrum disorder or other psychiatric disorders. Data from this study will be used to recommend pediatric doses that result in comparable exposures to those observed in currently approved adult doses of Latuda® (40, 80, 120 and 160 mg/day) in subsequent efficacy and safety studies.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must provide written informed consent, if emancipated, written assent and be willing to participate in the study. Written informed consent from parent(s) or legal guardian(s) with sufficient intellectual capacity to understand the study and support subjects' adherence to the study procedures must be obtained for subjects who are not emancipated.
* Male or female subjects 6 to 17 years of age, inclusive. Subject must be 17 years or less at the follow-up visit.
* Subject is judged by the investigator to be clinically stable (ie, no psychiatric hospitalization within the past 12 weeks; no imminent risk of suicide or injury to self, others or property; no recent addition, or change in dosage, of psychotropic medication intended for the treatment of the primary psychiatric condition in the past 4 weeks) but symptomatic (ie, some active symptoms of the primary psychiatric condition are present for which an atypical antipsychotic agent is judged to be an acceptable treatment option).
* Subjects with the following diagnoses will be eligible for participation: primary schizophrenia spectrum diagnosis (schizophrenia, schizoaffective, schizophreniform or psychotic disorder Not Otherwise Specified (NOS), bipolar spectrum disorder (bipolar I, II or bipolar NOS), pervasive developmental disorder (PDD) including autistic spectrum disorder (autistic disorder, Asperger's syndrome, or Pervasive Developmental Disorder-Not Otherwise Specified (PDD-NOS), attention-deficit hyperactivity (ADHD) with aggressive behavior [meeting co-morbid diagnostic criteria for Conduct Disorder/Disruptive Behavior Disorders Not Otherwise Specified (CD/DBD NOS), or Tourette's syndrome, via clinical interview (using MINI-Kid plus diagnostic interview and the Diagnostic and Statistical Manual of Mental Disorders, 4th edition Text Revision (DSM-IV-TR) as a reference). Autistic disorder should also be confirmed by the Autism Diagnostic Interview, Revised (ADI-R).
* Within 5th to 95th percentile for gender specific weight-for-age and height-for-age Growth Charts from National Center for Health Statistics.
* No clinically relevant abnormal laboratory values.
* No clinically relevant abnormal vital sign values/findings.
* Females who participate in this study:
* are unable to become pregnant (eg, premenarchal, surgically sterile etc) -OR-
* are willing to remain sexually abstinent (not engage in sexual intercourse) from Day 1 to 30 days after discharge on Day 11; -OR-
* are sexually active and willing to use an effective method of birth control (eg, male using condom and female using condom, diaphragm, contraceptive sponge, spermicide, contraceptive pill, or intrauterine device) from Day -1 to 30 days after discharge on Day 11.
* Males must be willing to remain sexually abstinent or use an effective method of birth control (eg, condom) from Day -1 to 30 days after discharge on Day 11.
* Willing and able to remain off any antipsychotic medication other than lurasidone for the duration of the study, if, in the investigator's opinion the subject is not at risk for worsening symptoms.
* Willing and able to swallow the size and number of lurasidone tablets specified per protocol.
* Willing and able to adhere to protocol-specified meal requirements during dosing.
* Have a stable living arrangement for at least 3 months prior to Day -1 and agrees to return to a similar living arrangement after discharge on Day 11. Homeless subjects may not be enrolled.

Exclusion Criteria:

* Clinically significant neurological, metabolic (including type 1 diabetes), hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, carcinoma, and/or urological disorder such as unstable angina, congestive heart failure (uncontrolled), or central nervous system (CNS) infection that would pose a risk to the subjects if they were to participate in the study or that might confound the results of the study.
* Note: Active medical conditions that are minor or well-controlled are not exclusionary if they do not affect risk to the subject or the study results. In cases in which the impact of the condition upon risk to the subject or study results is unclear, the Medical Monitor should be consulted. Any subject with a known cardiovascular disease or condition (even if under control) must be discussed with the Medical Monitor before being enrolled to the study.
* Evidence of any chronic organic disease of the CNS such as tumors, inflammation, active seizure disorder, vascular disorder, Parkinson's disease, or other forms of dementia, myasthenia gravis, or other degenerative processes. In addition, subjects must not have a history of mental retardation or persistent neurological symptoms attributable to serious head injury. Past history of febrile seizure, drug-induced seizure, or alcohol withdrawal seizure is not exclusionary.
* Known presence or history of hepatic insufficiency or subject's estimated creatinine clearance is < 80 mL/min/1.73 m2 by the following Bedside Schwartz equation for use with creatinine methods with calibration traceable to isotope dilution mass spectrometry (IDMS): Creatinine clearance (mL/min/1.73 m2) = (0.41 height) / serum creatinine concentration, where height in cm and serum creatinine in mg/dL.
* Clinically significant finding(s) on physical examination determined by the investigator to pose a health concern to the subject while on study.
* A history or presence of abnormal ECG, which in the investigator's opinion is clinically significant. Screening ECGs will be centrally over-read, and eligibility will be determined based on the over-read.
* Known history or presence of clinically significant intolerance to any antipsychotic medications including but not limited to angioedema, serotonin or neuroleptic malignant syndromes, moderate to severe dystonia, or moderate to severe tardive dyskinesia.
* Clinically significant alcohol abuse/dependence or drug abuse/dependence based on MINI-Kid criteria within the last 6 months prior to screening.
* Clinically significant orthostatic hypotension (ie, a drop in systolic blood pressure of 20 mmHg or more and/or drop in diastolic blood pressure of 10 mmHg or more within 3 minutes of standing up).
* Presence or history (within the last year) of a medical or surgical condition (eg, gastrointestinal disease) that might interfere with the absorption, metabolism, or excretion of orally administered lurasidone.
* Positive breath alcohol test at screening or on Day -1.
* Positive test results at screening or on Day -1 for:
* Urine drugs of abuse (amphetamines, barbiturates, benzodiazepines, cocaine, opiates, phencyclidine, cannabinoids, and methadone). However, a positive test for amphetamines, barbiturates, opiates, benzodiazepines or methadone may not result in exclusion of subjects if the investigator determines that the positive test is as a result of prescription medicine(s).
* Pregnancy test (only in female subjects ≥ 8 years old).
* Lifetime history of human immunodeficiency virus (HIV) positive or acquired immune deficiency syndrome (AIDS), or history of Hepatitis B or C, or a positive test for Hepatitis B or C at screening (for subjects without a history).
* Participated in another clinical trial or receiving an investigational product within 30 days prior to study drug administration.
* Use of any inhibitor or inducer of CYP3A4 taken within 28 days prior to drug administration and until discharge on Day 11. Exceptions (eg, for grapefruit juice consumption) may be discussed on a case-by-case basis with the medical monitor.
* Use of concomitant medications that consistently prolong the QT/QTc interval within 28 days prior to Day -1 to follow-up.
* Received depot neuroleptics unless the last injection was at least 1 month or 1 treatment cycle prior to Screening, whichever is longer.
* Received treatment with antidepressants within 3 days, fluoxetine or olanzapine plus fluoxetine combination within 28 days, MAO inhibitors within 14 days prior to Day -1 to follow-up.
* Use of any antipsychotic medication (other than study drug), carbamazepine, oxcarbazepine or fluvoxamine, within 3 days prior to Day -1 (7 days prior to Day -1 for aripiprazole) and until follow-up.
* Does not tolerate venipuncture or has any bleeding disorder that would complicate blood drawing.
* Females who are pregnant, lactating, or likely to become pregnant during the study.
* Donation or loss of whole blood within 60 days prior to drug administration.
* Has a prolactin concentration greater than or equal to 100 ng/mL at screening.
* Unwilling to abstain from vigorous exercise from Days -1 to 1 and from Days 9 to 10.
* Subject answers "yes" to "Suicidal Ideation" Items 4 or 5 on the C-SSRS.
* Subject is considered by the investigator to be at imminent risk of suicide or injury to self, others, or property during the study. Subject has a history of one or more serious suicide attempts (based on the investigator's judgment) in the 12 months prior to screening. Subjects determined to be at risk of suicide or injury, as assessed by the investigator at screening, will be referred for further psychiatric evaluation.
* Clinically relevant history of drug hypersensitivity to lurasidone or any components in the formulation.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 105 (Actual)
Dates: Start 2012-06; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lurasidone Medical Director, Study Director — Sumitomo Pharma America, Inc.
Locations (10):
- United States (10):
  - Woodland International Research Group, Inc., Little Rock, Arkansas
  - Woodland Northwest Research, LLC, Springdale, Arkansas
  - World Wide Research Centers Inc., Murrieta, California
  - Segal Institute for Clinical Research, Fort Lauderdale, Florida
  - Miami Children's Hospital, South Miami, Florida
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - University of Cincinnati, Dept. of Psychiatry & Behavioral Neuroscience, Cincinnati, Ohio
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - CRI Worldwide, LLC, Philadelphia, Pennsylvania
  - Aspen Clinical Research, Orem, Utah

REFERENCES:
- [Derived] Findling RL, Goldman R, Chiu YY, Silva R, Jin F, Pikalov A, Loebel A. Pharmacokinetics and Tolerability of Lurasidone in Children and Adolescents With Psychiatric Disorders. Clin Ther. 2015 Dec 1;37(12):2788-97. doi: 10.1016/j.clinthera.2015.11.001. Epub 2015 Nov 26. PMID 26631428

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Total subjects randomized was 105. Total subjects with PK data was 102.
Period: Overall Study
Arm/Group | Lurasidone Oral Tablets
Started | 105
Completed | 90
Not Completed | 15
Not completed — Adverse Event | 9
Not completed — Protocol Violation | 1
Not completed — Withdrawal by Subject | 1
Not completed — Did not comply with Study Produre | 1
Not completed — Family emergency | 1
Not completed — Per Sponsor Decision | 2

BASELINE CHARACTERISTICS:
Arm/Group | Lurasidone Oral Tablets
Number analyzed (Participants) | 105
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 105
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37
  Male | 68
Race/Ethnicity, Customized [Number; unit: participants]
  Black or African American | 23
  White | 82
Region of Enrollment [Number; unit: participants]
  United States | 105

OUTCOME MEASURES:

1. Primary Outcome: Lurasidone Primary Pharmacokinetic Parameters
Description: Lurasidone AUClast (Day 1) and AUC0-∞ (Day 1) AUC0-24 (Day 10 or Day 12)
Time Frame: Day 1 - pre-dose, 30 minutes, 1 hour, 2 hours, 4 hours, 6 hours, 8 hours, 12 hours, 24 hours, and 48 hours. Day 10/12: 30 minutes, 1 hour, 2 hours, 4 hours, 6 hours, 8 hours, 12 hours, 24 hours
Population: Participants for PK analysis included all subjects who received at least 1 dose of study drug and had at least 1 measured concentration at a scheduled PK timepoint after start of dosing for at least 1 PK analyte.
  For some PK parameters, some subjects didn't have PK data.
Measure: Mean (Standard Deviation); unit: ng.h/mL
Arm/Group | Lurasidone Oral Tablets
Number analyzed (Participants) | 102
ng.h/mL
  AUC last (ng.h/mL) -Day 1 20 mg n=16 | 78 (44.9)
  AUC last (ng.h/mL) -Day 1 40 mg n=24 | 140 (65.4)
  AUC last (ng.h/mL) -Day 1 80 mg n=54 | 300 (140)
  AUC0-24 (ng.h/mL) -D 10/12 20 mg n=16 | 115 (72.2)
  AUC0-24 (ng.h/mL) -D10/12 40 mg n=21 | 154 (67.4)
  AUC0-24 (ng.h/mL) -D10/12 80 mg n=17 | 387 (194)
  AUC0-24 (ng.h/mL) -D10/12 120 mg n=16 | 494 (271)
  AUC0-24 (ng.h/mL) -D 10/12 160 mg n=13 | 590 (227)
  AUC0-∞(ng.h/mL) -D 1 20 mg n=16 | 83.8 (48.3)
  AUC0-∞(ng.h/mL) -D 1 40 mg n=19 | 153 (69.8)
  AUC0-∞(ng.h/mL) -D 1 80 mg n=50 | 328 (163)

2. Primary Outcome: Lurasidone Peak Serum Concentration (Cmax)
Description: Cmax will be listed and summarized in tabular format
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Lurasidone Oral Tablets
Number analyzed (Participants) | 102
ng/mL
  Cmax (ng/mL)-Day 1 20 mg n=16 | 24.4 (14.1)
  Cmax (ng/mL)-Day 1 40 mg n=24 | 38.3 (22.4)
  Cmax (ng/mL)-Day 1 80 mg n=55 | 68.2 (37.5)
  Cmax (ng/mL)-D10/12 20 mg n=16 | 30 (18)
  Cmax (ng/mL)-D10/12 40 mg n=21 | 36.2 (17.5)
  Cmax (ng/mL)-D10/12 80 mg n=17 | 80 (59.6)
  Cmax (ng/mL)-D10/12 120 mg n=16 | 94.2 (46.6)
  Cmax (ng/mL)-D10/12 160 mg n=13 | 99.7 (44.3)

3. Secondary Outcome: Number of Participants With Serious Adverse Events and Non-serious Adverse Events
Description: Serious adverse event and adverse events data will be listed and summarized as per MedDRA V15.0
Time Frame: 11 Days
Measure: Number; unit: participants
Arm/Group | Lurasidone Oral Tablets
Number analyzed (Participants) | 105
participants | 105

ADVERSE EVENTS:
Time Frame: June 19, 2012 through May 6, 2013
Arm/Group | Lurasidone Oral Tablets
Serious Adverse Events (participants affected / at risk) | 2/105
Other Adverse Events (participants affected / at risk) | 76/105
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lurasidone Oral Tablets (N=105)
Parkinsonism (Nervous system disorders) | 1 (1)
Dystonia (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lurasidone Oral Tablets (N=105)
Nausea (Gastrointestinal disorders) | 18 (20)
Vomiting (Gastrointestinal disorders) | 16 (18)
Upper Abdominal Pain (Gastrointestinal disorders) | 6 (6)
Somnelence (Nervous system disorders) | 44 (104)
Sedation (Nervous system disorders) | 19 (35)
Dystonia (Nervous system disorders) | 5 (7)
Dyskinesia (Nervous system disorders) | 5 (5)
Anxiety (Psychiatric disorders) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In addition to the <60-180 day restriction above, since this is a multicenter study, 1st publication of study results shall be made with other participating study sites as a multicenter publication; provided, if a multicenter publication is not forthcoming within 24 months following completion of study at all sites, the PI shall be free to publish.